CLINICAL TRIAL: NCT07070518
Title: An Open-Label Phase 1/2A Study of GV20-0251 in Participants With Advanced and/or Refractory Solid Tumor Malignancies
Brief Title: Study of GV20-0251 in Participants With Solid Tumor Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GV20 Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GV20-0251-300
Record Dates: First submitted 2025-06-26; First posted 2025-07-17 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor Cancer; Adult Refractory Cancer; Endometrial Carcinoma (EC); Squamous Head and Neck Carcinoma; pMMR/MSS Adenocarcinoma of the Colon or Rectum; Non-Small Cell Lung Cancer; Melanoma; HCC - Hepatocellular Carcinoma; Small Cell Lung Cancer
MeSH Terms: conditions — Neoplasms; Endometrial Neoplasms; Carcinoma, Non-Small-Cell Lung; Melanoma; Carcinoma, Hepatocellular; Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GV20-0251 (Experimental)
  Interventions: Drug: GV20-0251

INTERVENTIONS:
Drug: GV20-0251 — Part A: Increasing doses of GV20-0251 administered by intravenous (IV) infusion once every 3 weeks Part B: GV20-0251 preliminary RP2D administered by IV infusion once every 3 weeks

SUMMARY:
This is a Phase 1 and Phase 2 study of GV20-0251 being developed for the treatment of participants with advanced solid tumors, who are refractory to approved therapies or other standard of care.

DETAILED DESCRIPTION:
This is a Phase 1/2A non-randomized, open-label, multi-center study to be conducted in 2 parts (A and B).

Part A is a safety run-in portion. A 3+3 dose escalation scheme will be used to evaluate the safety and tolerability of GV20-0251, and to establish the maximum tolerated dose (MTD) or the preliminary recommended Phase 2 dose (RP2D).

In Part B, the Simon 2-stage design will be utilized to further characterize the anti-tumor activities, safety, tolerability, pharmacokinetics, and pharmacodynamics of GV20-0251 at the preliminary RP2D across multiple expansion cohorts involving eligible participants.

ELIGIBILITY:
Inclusion Criteria:

* Before conducting any study-specific procedures, voluntarily sign an informed consent form.
* Be able and willing to participate throughout the entire study period and comply with study procedures.
* participants ≥18 years of age
* Previously treated, histologically-confirmed advanced solid malignancy with progressive disease requiring therapy (Refractory or intolerant to standard therapies, must have received the standard of care therapy)
* Participants must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST version 1.1)
* For participants who have received prior treatment with a checkpoint inhibitor there must be documented disease progression
* ECOG performance status of 0 or 1 before C1D1
* Part B Participants must be willing to provide fresh tumor biopsy (core biopsy) both pre-treatment and on-treatment, if clinically feasible
* Disease-free of active second/secondary or prior malignancies for ≥ 2 years Laboratory test results within the required parameters
* Women of childbearing potential (WOCBP) and men must agree to use adequate contraception

Exclusion Criteria:

* Participants with acute leukemia or CLL
* Participant with heart disease (NYHA ≥ Level II), myocardial infarction within the past 6 months, or unstable arrhythmia
* Fridericia-corrected QT interval (QTcF) > 470 msec, or the presence of congenital long QT syndrome, or a history of clinically significant electrocardiogram (ECG) abnormalities (including pericarditis) that, in the investigator's judgment, may affect the subject's safety.
* Active, uncontrolled bacterial, viral, or fungal infections requiring systemic therapy within 7 days before C1D1
* Participant has active autoimmune disease or other medical conditions requiring chronic systemic steroid or immunosuppressive therapy
* Known human immunodeficiency virus (HIV) infection, known hepatitis B virus (HBV), or hepatitis C virus (HCV) infection, unless meeting the specific conditions.
* History of major organ transplant and/or a bone marrow transplant
* Symptomatic central nervous system (CNS) malignancy or metastasis
* Serious nonmalignant disease
* Pregnant or nursing women
* Major surgery within 28 days prior to the first dose of study medication
* Prior anticancer therapy within 4 weeks or 5 half-lives (whichever is shorter) before the first dose of GV20-0251 on Cycle 1 Day 1 (C1D1), with the exceptions.
* History of severe allergic reactions to biologic therapy, which in the investigator's judgment may increase the subject's risk.
* Radiation therapy for symptomatic lesions within 14 days prior to C1D1 dosing.
* Active substance abuse
* Any history of an immune-related ≥ Grade 3 AE attributed to prior cancer immunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2027-07-16 (Estimated); Study Completion 2028-09-16 (Estimated)

PRIMARY OUTCOMES:
Evaluate anti-tumor activities with GV20-0251 | From Cycle 1 Day 1 dosing (each cycle is 21 days) until disease progression or end of study (whichever occurs first, up to 24 months)
  Objective Response Rate (ORR) assessed by RECIST v1.1 (Response Evaluation Criteria in Solid Tumors, Version 1.1)

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Li Y, Wu X, Sheng C, Liu H, Liu H, Tang Y, Liu C, Ding Q, Xie B, Xiao X, Zheng R, Yu Q, Guo Z, Ma J, Wang J, Gao J, Tian M, Wang W, Zhou J, Jiang L, Gu M, Shi S, Paull M, Yang G, Yang W, Landau S, Bao X, Hu X, Liu XS, Xiao T. IGSF8 is an innate immune checkpoint and cancer immunotherapy target. Cell. 2024 May 23;187(11):2703-2716.e23. doi: 10.1016/j.cell.2024.03.039. Epub 2024 Apr 23. PMID 38657602